CLINICAL TRIAL: NCT01210937
Title: Early Warning and Optimization Strategy in Carotid Endarterectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Liu Chang-wei, Vascular Surgery, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pumch-CAS
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2010-09

CONDITIONS: Carotid Stenosis; Carotid Artery Diseases; Stroke; Vascular Diseases
Keywords: Internal Carotid Artery Stenosis; Carotid Endarterectomy; Stroke; Cerebrovascular; Atherosclerosis
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases; Stroke; Vascular Diseases; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CEA and TCD monitoring (Experimental): CEA involves a neck incision and physical removal of the plaque from the inside of the artery.During the surgery, the patient will be monitored by TCD.
  Interventions: Procedure: CEA and TCD monitoring

INTERVENTIONS:
Procedure: CEA and TCD monitoring — All patients will receive carotid endarterectomy. During the surgery, all of them will be monitored by TCD. Record the blood flow velocity and blood pressure on specified time.

SUMMARY:
Carotid endarterectomy has been proven effective in prevention of cerebral vascular events in patients with severe carotid artery stenosis (symptomatic,>50%;asymptomatic,60%). But during the surgery, when the carotid artery is clipping, the patient will have the chance to have hypoperfusion or stroke. Our study is designed to determine how to use TCD to reduce the risk of death and nonfatal stroke in patients .

DETAILED DESCRIPTION:
AHA guidelines recommend carotid endarterectomy (CEA) for severe carotid stenosis. But during CEA, there is little chance that the patient suffer from severe hypoperfusion or stroke. So we use TCD to monitor the blood flow of brain in the surgery and keep the blood pressure stable. The sudy is designed to find out whether the index which we found in previous work is more sensitive to show the blood flow of middle cerebral artery.

ELIGIBILITY:
Inclusion Criteria:

* Carotid artery stenosis detectable by duplex ultrasound, and no previous procedure done on it, which might well need procedural treatment now with CEA or CAS.
* Already started any appropriate medical treatment (eg, statin, aspirin etc), and already recovered from any necessary coronary procedures (eg, CABG)
* Patient seems fit and willing for follow-up in person (at 1 month) and by annual letter (for at least 5 years)
* Some type of angiography (eg, MRA or CTA) has already been done that has shown that CEA .

Exclusion Criteria:

* Small likelihood of worthwhile benefit (eg, very low risk of stroke because stenosis is very minor, or major co-morbidity or life-threatening disease, such as advanced cancer)

Ages: 40 Months to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  The number of death during the first month after procedure, no matter whether the cause of death is related to the procedure

SECONDARY OUTCOMES:
cardiac and neurological morbidity (TIA and CVA) | 12 months
brain hyperperfusion | 12 months
long term recurrence | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Liu Changwei, bachelor, Study Chair; Liu Bao, doctor, Principal Investigator
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- See also: the website of the vascular surgery department of PUMCH — http://www.vascular.cn/